CLINICAL TRIAL: NCT04066543
Title: A Single-center Randomized Controlled Clinical Trial of TACE Combined With Anlotinib Comparing With TACE in the Treatment of Middle-advanced Hepatocellular Carcinoma (HCC) Patients
Brief Title: TACE Combined With Anlotinib Treatment of Middle-advanced Hepatocellular Carcinoma (HCC) Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTNZJ-002
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — anlotinib

STUDY DESIGN:
Intervention Model Description: TACE vs.TACE+Anlotinib
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TACE group (Active Comparator): Device: Transcatheter arterial chemoembolization(TACE)
  Interventions: Device: TACE
- TACE+Anlotinib group (Experimental): Device: Transcatheter arterial chemoembolization Drug: Anlotinib Anlotinib hydrochloride capsule, according to the recommended dose, po, qd, continuous oral 2 weeks stop for 1 week, 3 weeks for a cycle.
  Interventions: Device: TACE; Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Device: TACE — The modified Seldinger puncture was used to puncture the cutaneous-femoral artery, insert the catheter and perform hepatic artery angiography. The location, morphology and blood supply of liver tissue lesions were comprehensively understood. The use of chemotherapeutic drugs and the dosage of iodized oil as the embolic agent were determined according to the general situation. The catheter was injected into the supply vessel of the tumor, and 5-FU and adriamycin were injected according to the situation. The embolic agent was injected with iodized oil as carrier, mixed with chemotherapeutic drugs at the same time, and then assisted with gelatin sponge for embolization. Antiemetic drugs were given before treatment and hepatoprotective drugs were given after operation. Until the disease progresses.
Drug: Anlotinib Hydrochloride — Anlotinib hydrochloride capsule, according to the recommended dose, po, qd, continuous oral 2 weeks stop for 1 week, 3 weeks for a cycle.
  Other Names: Anlotinib
  Arms: TACE+Anlotinib group

SUMMARY:
This study was designed to evaluate the effectiveness of Anlotinib in middle-advanced Hepatocellular Carcinoma (HCC) Patients.

DETAILED DESCRIPTION:
The aim of this study is to include 40 patients with middle-advanced Hepatocellular Carcinoma .These patients were randomly allocated to TACE treatment group or TACE+Anlotinib treatment group.The treatment effectiveness, local tumor control and survival outcome between the two groups were compared.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has no contraindication to chemotherapy, and has no obvious obstacles in the function of major organs such as heart, lung, liver and kidney;
2. Subject has middle-advanced liver cancer of Barcelona Clinic Liver Cancer stages B/C ;
3. Liver function child-pugh class A or B; Karnofsky (KPS) score > 60 points;
4. Subject could not accept surgical resection or refuse surgical operation;and who did not receive other treatment before operation.

5.18~75 years old; ECOG PS score: 0-1 points; expected survival period is more than 3 months.

Exclusion Criteria:

1. Subject has contraindications to chemotherapy;
2. Subject has obstacle in the function of major organs such as heart, lung, liver and kidney;
3. Severe coagulation dysfunction (prothrombin time > 18 s or hemorrhagic tendency);
4. Uncontrollable hypertension and portal hypertension;
5. Hepatic artery-portal vein or hepatic vein fistula or portal vein trunk cancer thrombus;
6. A large amount of ascites or refractory ascites;
7. With distant metastasis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-30 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 12 months
  Progress Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Shao, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang D, Zhang Z, Luo J, Zheng J, Mao X, Tsilimigras DI, Chun HJ, Zeng H. Efficacy and safety of transarterial chemoembolization alone compared to its combination with anlotinib among patients with intermediate or advanced stage hepatocellular carcinoma: a phase II randomized controlled trial. J Gastrointest Oncol. 2024 Aug 31;15(4):1627-1635. doi: 10.21037/jgo-24-497. Epub 2024 Aug 28. PMID 39279973